CLINICAL TRIAL: NCT06804915
Title: A Mobile App For Drug Dosage Calculation In The Context Of Pediatric And Adult Resuscitation: A Cross-Over Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Matthieu Vincent, Emergency medicine and Pediatric emergency medicine specialist, Université de Sherbrooke
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-922
Record Dates: First submitted 2025-01-10; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Mobile App Use in Resuscitation
Keywords: mobile app; smartphone; resuscitation; drug errors

STUDY DESIGN:
Intervention Model Description: Each team will conduct one adult and one pediatric resuscitation scenario using the EZResus application, along with one adult and one pediatric resuscitation scenario following standard protocols.The teams will be individually randomized to start the scenarios either with or without the medical application using sealed envelopes. Standard protocol is defined as standard care using any resources usually used by professionals, except for medical calculator applications.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medical calculator application use (EzResus) (Experimental): Participants (physicians and nurses) will be allowed to use a medical calculator application called EzResus. They will receive a 5-minute training prior to the simulations. Participants are also allowed to use other ressources, such as local protocols, medication administration guide.
  Interventions: Behavioral: simulation
- Standard care (Active Comparator): Participants are also allowed to use the ressources they use in their practice, apart from a medical calculator application. They are allowed to use local protocols, medication administration guides, medical mobile apps that don't calculate drug doses.
  Interventions: Behavioral: simulation

INTERVENTIONS:
Behavioral: simulation — Each team of physician and nurses will participate in 4 scenarios: 2 adult, 2 pediatric. In each scenario, physician and nurses will have a clinical description of the scenario with the age and weight of each patient.
  The simulations will be conducted at the clinical simulation laboratory at Jean-Marc Lepage Pavilion of the University of Sherbrooke using high-fidelity mannequins. SimMan 3GPus will be used for adult scenarios and SimJunior for pediatric scenarios, both from Laerdal company. Participants will receive a briefing containing key information about the scenario and the patient just before starting the simulation.
  During the scenarios, the physician is expected to prescribe medications by mentioning the name, the dose and the route of administration of every medication. Moreover, if multiple dilution for a medication is possible, the physician is expected to mention the desired dilution.

SUMMARY:
The purpose of this study is to investigate whether the use of the EZResus app by physicians and nurses reduces medication errors in simulated adult and pediatric resuscitation scenarios compared to the use of standard protocols. This study is a randomized controlled crossover trial with two groups comparing the use of EZResus app with standard protocol in four simulated resuscitation scenarios. The participants will form resuscitation teams, each including an attending physician and two nurses responsible for the preparation and administration of medications. Each team will conduct one adult and one pediatric resuscitation scenario using the EZResus application, along with one adult and one pediatric resuscitation scenario following standard protocols.The teams will be individually randomized to start the scenarios either with or without the medical application using sealed envelopes. The participants will be recruited from one regional hospital (Haut-Richelieu hospital) and one university hospital (Charles LeMoyne Hospital).

DETAILED DESCRIPTION:
The simulations will be conducted at the clinical simulation laboratory at Jean-Marc Lepage Pavilion of the University of Sherbrooke using high-fidelity mannequins. During the scenarios, the physician is expected to prescribe medications by mentioning the name, the dose and the route of administration of every medication. Moreover, if multiple dilution for a medication is possible, the physician is expected to mention the desired dilution.

The first pediatric scenario will be a refractory status epilepticus situation where we will evaluate the dosing of benzodiazepines, followed by a 2nd line antiepileptic agent (levetiracetam or phenytoin). If asked, the patient will have hypoglycemia and need IV glucose. The patient will eventually require intubation where we will evaluate the dosage of the induction agent, neuromuscular blocking agent (NMBA), ventilation parameters and intubation equipment (laryngoscope blade and endotracheal tube size). Post intubation, the participant will need to start a perfusion for refractory status epilepticus (midazolam or propofol).

The second pediatric scenario will be a cardiac arrest. The patient will be in ventricular fibrillation and we will evaluate the dosage of epinephrine, antiarrhythmic medication (amiodarone and/or lidocaine) and electric voltage for defibrillation. After return to spontaneous circulation, the patient will require vasopressors (epinephrine perfusion) for hypotension, following PALS guidelines.

The first adult scenario will be a case of calcium channel-blocker toxicity where we will evaluate the dosing of activated charcoal followed by high-dose insulin, dextrose and calcium. The patient will deteriorate and need a vasopressor perfusion and will eventually need intubation where we will evaluate the induction agent, NMBA, ventilation parameters and intubation equipment (laryngoscope blade and endotracheal tube size).

The second adult scenario will be an aortic dissection. We will evaluate the dose of beta blocker (labetalol or esmolol) and the dose of clevidipine, nicardipine or nitroprusside. We will also evaluate the dosage of fentanyl for analgesia.

ELIGIBILITY:
Inclusion Criteria: The participants will be recruited from one regional hospital (Haut-Richelieu hospital) and one university hospital (Charles LeMoyne Hospital).

* Emergency physicians or emergency nurses working in the resuscitation room and working in one of the two eligible hospital centers.

Exclusion Criteria:

* Being part of the research team or affiliated in any way with the EZResus team.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Drug administration appropriate or not | duration of the simulation: 15-25 minutes per scenario
  In this study, the drug administration will be classified as either appropriate or inappropriate, with inappropriate administration being defined by one or more of the following criterias :
  * the administration of the incorrect medication
  * the use of an inappropriate route of administration
  * a prescribed dosage that deviates by more than 10% from the appropriate dose (as defined in the medication tables in appendix) or
  * an administered dosage that deviates by more than 10% from the prescribed dosage
  * The omission of a medication considered essential for treatment.

SECONDARY OUTCOMES:
Drug administration appropriate or not - prescription phase | duration of the simulation: 15-25 minutes per scenario
  As defined for the primary outcome measure, error occurring during the prescription, either from a verbal prescription or written prescription
Drug administration appropriate or not | duration of the simulation: 15-25 minutes per scenario
  As defined for the primary outcome measure. Error occurring during the administration phase.
time to drug prescription | duration of the simulation: 15-25 minutes per scenario
  measured from the beginning of the scenario to the physician's verbal prescription (defined as the first mention of the drug's name)
time for drug preparation | duration of the simulation: 15-25 minutes per scenario
  measured from the physician's verbal prescription to the start of drug preparation by the nurse
time to drug delivery | duration of the simulation: 15-25 minutes per scenario
  measured from the verbal prescription to the beginning of administration of the drug
mental workload | The questionnaire will be administered twice: once after completing two scenarios without the application and once after completing two scenarios with the application
  will be assessed using the simplified NASA Task Load Index method, which employs a questionnaire featuring five 7-point scales, rating performance across six dimensions: mental demand, physical demand, temporal demand, effort, performance and frustration level.
Deviation in endotracheal size | duration of the simulation: 15-25 minutes per scenario
  In some scenarios, whenever a pediatric simulated patient is intubated.
Deviation in laryngoscope blade sizes | duration of the simulation: 15-25 minutes per scenario
  Apply to the 2 pediatric scenarios
Electrical voltage for defibrillation | duration of the simulation: 15-25 minutes per scenario
  Electrical voltage for defibrillation - whether accurate or innacurrate
Ventilatory parameters appropriateness | duration of the simulation: 15-25 minutes per scenario
  appropriateness of volumes and respiratory rates

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Charles-Le Moyne, Greenfield Park, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
all requested data